CLINICAL TRIAL: NCT04255316
Title: Modified Method of Eversion Carotid Endarterectomy in Patients With Extensive Atherosclerotic Disease of Carotid Bifurcation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-01

CONDITIONS: Carotid Stenosis; Carotid Artery Diseases
Keywords: carotid endarterectomy; eversion carotid endarterectomy; prophylaxis of ischemic stroke; carotid arteriosclerosis; carotid artery plasty
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified eversion (Experimental): Patients with extensive atherosclerotic lesion of the carotid bifurcation (more 25mm in internal carotid artery) undergo a modified eversion carotid endarterectomy
  Interventions: Procedure: Modified method of eversion carotid endarterectomy
- Standard eversion (Active Comparator): Patients with extensive atherosclerotic lesion of the carotid bifurcation (more 25mm in internal carotid artery) undergo a standard eversion carotid endarterectomy
  Interventions: Procedure: Standard method of eversion carotid endarterectomy

INTERVENTIONS:
Procedure: Modified method of eversion carotid endarterectomy — Mini approach for CCA bifurcation - Clamping ICA, ECA and CCA - ICA is cut off with a scalpel at the mouth itself - Dissection of the ICA and ECA in the distal direction to the distal border of the atherosclerotic plaque - Endarterectomy - Performing of a new bifurcation of the CCA with prolene 7/0
  Arms: Modified eversion
Procedure: Standard method of eversion carotid endarterectomy — standard eversion technic
  Arms: Standard eversion

SUMMARY:
A prospective comparative randomized single-centre non-inferiority trial. The purpose of this study is to compares of modified method of eversion carotid endarterectomy with standard eversion carotid endarterectomy for 3,6 and 12 months days after operation in patients with extensive atherosclerotic disease of carotid bifurcation

DETAILED DESCRIPTION:
Introduction. Performing eversion endarterectomy some difficulties arise. Firstly, it requires a great deal of coherence between the work of the surgeon and the first assistant, as well as a great experience of the latter. Secondly, in some cases, there are difficulties in visualizing the distal margin of the intima: in the absence of a rigid skeleton, the soft unchanged artery walls after removal of the plaque subside, making it difficult to visualize possible fragments of the intima. Thirdly, the cost of the error is high: with a random de-version, repeated eversion turns out to be impossible. It should be noted that the use of an eversion technique becomes difficult to implement, and sometimes impossible, with extended stenosis, since a very high allocation of the ICA is required, which increases the invasiveness of the operation and the difficulty of access. With prolonged stenosis, the carotid endarterectomy remains the option of choice. The modification used eversion carotid endarterectomy combines the advantages of both methods, and also eliminates the limitations of the carotid endarterectomy and eversion carotid endarterectomy.

The aim of study. The purpose of this study is to compares of modified method of eversion carotid endarterectomy with standard eversion carotid endarterectomy for 3,6 and 12 months days after operation in patients with extensive atherosclerotic disease of carotid bifurcation

ELIGIBILITY:
Inclusion Criteria:

* patients with stenosis of ICA 70-99% (ultrasound - NASCET and CT angiography)
* patients with a extensive lesion of the ICA (plaque < 2 cm) by ultrasound - NASCET and CT angiography

Exclusion Criteria:

* patients with a extensive lesion of the ICA (plaque < 2 cm),
* patients with a contralateral occlusion of the ICA
* patients with stroke in ischemic type in the acute period.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Assessment of total stroke rate | 30 days
  assessment of the total stroke rate in patients undergoing intervention after 30 days
Assessment of mortality rate | 30 days
  assessment of the mortality rate in patients undergoing intervention after 30 days

SECONDARY OUTCOMES:
Assessment of stroke frequency | 12 months
  assessment of stroke frequency in patients undergoing intervention after 12 months
Assessment of the incidence of internal carotid artery restenosis | 3, 6, 12 months
  Assessment of the incidence of internal carotid artery restenosis after 3, 6 and 12 months

OTHER OUTCOMES:
Evaluation of speed flow in carotid bifurcation by ultrasound duplex scan | 24 hours, 30 days, 3, 6 and 12 months
  Evaluation of speed flow, peak systolic velocity (cm/s) in common carotid artery, internal carotid artery and external carotid artery and their ratios using ultrasound duplex scan.

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly Virgansky, MD, Principal Investigator — The Federal Budget-Funded Institution National Medical Surgical Center named after N. I. Pirogov
Locations (1):
- The Federal Budget-Funded Institution National Medical Surgical Center named after N. I. Pirogov of the Ministry of health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No